CLINICAL TRIAL: NCT01964235
Title: A Randomized Phase II, Double-blind, Placebo-controlled, Multi-center Study to Evaluate the Efficacy and Safety of INC280 in Adult Patients With Advanced Hepatocellular Carcinoma After Progression or Intolerance to Sorafenib Treatment
Brief Title: Study of Efficacy and Safety INC280 in Patients With Advanced Hepatocellular Carcinoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was cancelled by Sponsor.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CINC280X2203
Record Dates: First submitted 2013-10-14; First posted 2013-10-17 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: INC280, advanced hepatocellular carcinoma, c-MET pathway dysregulation.
MeSH Terms: interventions — capmatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- INC280 plus best supportive care (Experimental): Approximately 46 patients will be treated with INC280 600 mg twice a day plus best supportive care.
  Interventions: Drug: INC280
- Placebo plus best supportive care (Placebo Comparator): Approximately 23 patients will be treated with matching placebo twice a day plus best supportive care.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: INC280 — INC280 will be administered orally and continuously on a twice a day dosing schedule.
  Arms: INC280 plus best supportive care
Drug: Placebo — Placebo will be administered orally and continuously on a twice a day dosing schedule.
  Arms: Placebo plus best supportive care

SUMMARY:
This study is establish whether INC280 is safe and has beneficial effects in patients with advanced hepatocellular carcinoma known to have dysregulation of c-MET pathway and whose disease progressed while on, or after, treatment with sorafenib or who are intolerant to sorafenib.

Patients will be randomized in a 2:1 ratio to receive INC280 at 600mg BID plus best supportive care (BSC) or placebo plus BSC, until disease progression or intolerable to study treatment. Patients treated with placebo plus BSC will have the opportunity to receive INC280 treatment upon documented further disease progression (RECIST 1.1) per investigator's discretion after unblinding.

Patient will be stratified to geographical region (Asia vs Rest of World ) and tumor burden (present macroscopic vascular invasion and/or extra-hepatic spread vs not present).

DETAILED DESCRIPTION:
Study was cancelled by Sponsor prior to enrollment of patients.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed c-MET pathway dysregulation.- Hepatocellular carcinoma stage B or C according to the Barcelona Clinic Liver cancer staging classification. - Current cirrhotic status of Child-Pugh class A with no encephalopathy. - Documented disease progression during or after discontinuation of sorafenib treatment or intolerance to sorafenib treatment. - Measurable disease as determined by RECIST v1.1. - ECOG performance status ≤ 1

Exclusion Criteria:

* Previous local antineoplastic therapy or investigational drug completed less than 5 half-lives of the agent prior to randomization and have not recovered from clinically significant toxicity from such treatment to grade ≤1 by the NCI-CTCAE. - Received any targeted therapy other than sorafenib.
* Active bleeding within 28 days prior to screening visit including variceal bleeding (esophageal varices should be treated according to standard practice and procedure completed 28 days prior to screening visit). - Clinically significant venous or arterial thrombotic disease within past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12; Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Time to progression using Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1 | baseline, 6 weeks up to 6 months
  Time to progression is the time from the date of baseline evaluation to the date of the first documented radiological confirmation of disease progression.

SECONDARY OUTCOMES:
Best Overall Response | date of treatment, every 6 weeks up to 6 months
  Best overall response is defined as the best response recorded from the date of randomization until the date of last tumor assessment per RECIST version 1.1.
Overall Response Rate | baseline, every 6 weeks up to 6 months
  Overall Response Rate is defined as the proportion of patients with a best overall response of complete response or partial response at any time on study per RECIST version 1.1.
Disease Control Rate | baseline, every 6 weeks up to 6 months
  Disease control rate is defined as the proportion of patients with a best overall response of complete response, partial response or stable disease at any time on study per RECIST version 1.1.
Progression Free Survival | randomization, every 6 weeks up to 6 months
  Progression free survival is defined as the time from date of randomization to the date of the first radiologically documented progression or death due to any cause. If a patient has not experienced radiologically documented progression or death, progression free survival is censored at the date of last adequate tumor assessment.
Overall Survival | randomization until death, average 10 months
  Overall survival is defined as the time from date of randomization to the date of death due to any cause. If a patient is not known to have died, survival will be censored at the date of last contact.
Safety: adverse events, serious adverse events | From baseline until 30 days post study treatment
  Frequency, duration and severity of adverse events.
Safety: hematology and chemistry values, vital signs, electrocardiograms | From baseline until end of treatment, average 6 months from baseline
  Change from baseline values.
Tolerability of study drug | From date of randomization until end of treatment, average 6 months from baseline
  Tolerability will be assessed by summarizing the number of dose interruptions, dose reductions and dose intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (15):
- United States (2):
  - Massachusetts General Hospital Mass General Hospital, Boston, Massachusetts
  - Research Medical Center Onc Dept, Kansas City, Missouri
- Australia (2):
  - Novartis Investigative Site, Kogarah, New South Wales
  - Novartis Investigative Site, Heidelberg, Victoria
- France (4):
  - Novartis Investigative Site, Clichy
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nice
- Germany (2):
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Würzburg
- Hong Kong (2):
  - Novartis Investigative Site, Hong Kong
  - Novartis Investigative Site, Hong Kong SAR
- Novartis Investigative Site, Córdoba, Andalusia, Spain
- Switzerland (2):
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Geneva